CLINICAL TRIAL: NCT04985890
Title: A Proof of Concept Study to Evaluate the Safety and Efficacy of UB-421 in Combination With Chidamide for Reduction of HIV Reservoir as Compared to UB-421 Alone in ART Stabilized HIV-1 Patients Who Undergo ART Interruption
Brief Title: A Proof of Concept Study to Evaluate the Effect of UB-421 in Combination With Chidamide on HIV Viral Reservoir
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UBP Greater China (Shanghai) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UBP-A230-HIV
Record Dates: First submitted 2021-07-08; First posted 2021-08-02 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2022-08

CONDITIONS: HIV-1-infection
Keywords: UB-421; HIV
MeSH Terms: interventions — UB-421

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UB-421 monotherapy (Experimental): Subjects will receive 10 mg/kg UB-421 weekly infusion for 8 weeks.
  Interventions: Biological: UB-421
- UB-421 + chidamide combination therapy (Experimental): Subjects will receive 10 mg/kg UB-421 weekly infusion and 10 mg chidamide twice a week administration for 8weeks.
  Interventions: Other: UB-421+chidamide

INTERVENTIONS:
Biological: UB-421 — 10mg/kg weekly intravenous infusion to substitute for for antiretroviral therapy
  Arms: UB-421 monotherapy
Other: UB-421+chidamide — 10 mg/kg UB-421 weekly intravenous infusion to substitute for antiretroviral therapy, and combined with oral 10 mg chidamide twice a week for 8 weeks. Chidamide taken on the one day and three days after the administration of UB-421.
  Arms: UB-421 + chidamide combination therapy

SUMMARY:
* To assess the impact of UB-421 and chidamide in changing HIV-1 viral reservoir profile among HIV-1 suppressed patients who undergo short-term ART interruption.
* To evaluate the safety and tolerability of UB-421 combined with chidamide among HIV-1 suppressed patients who undergo short-term ART interruption.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible to be included in the study only if ALL of the following criteria apply:

1. HIV-1 sero-positive, with documented HIV-1 infection by official, signed, written history.
2. Male with body weight ≥ 50 kg or female with body weight ≥ 45 kg, aged 18 years or older.
3. Have been receiving at least (≧) 2 nucleoside/ nucleotide reverse transcriptase inhibitors (NRTI) plus one non-nucleoside reverse transcriptase inhibitor (NNRTI), protease inhibitor (PI, either boosted or un-boosted), integrase strand transfer inhibitor (INSTI) or entry inhibitor (EI) for more than 1 years.
4. Have more than 2 different alternative options of optimized ART regimen.
5. HIV-1 plasma viral load (VL) level well suppressed below 50 RNA copies/mL for at least (≧) 12 months.
6. No breastfeeding or pregnancy for women.
7. Both male and female patients and their partners of childbearing potential must agree to use 2 medically accepted methods of contraception (eg, barrier contraceptives [male condom, female condom, or diaphragm with a spermicidal gel], hormonal contraceptives [implants, injectable, combinational oral contraceptives, transdermal patches, or contraceptive rings], and intrauterine devices) during the course of the study (excluding women who are not of childbearing potential and men who have been sterilized). Females of childbearing potential must have a negative serum pregnancy test.
8. Subjects must sign the informed consent before undergoing any study procedures.

Exclusion Criteria:

Subjects meeting ANY of the following criteria will be excluded from the study:

1. Subjects with active systemic infections, except for HIV-1, that the investigator feels the infections may confound evaluation and treatment for HIV-1.
2. Any acquired AIDS-defining illness such as non-Hodgkin's lymphoma or Kaposi's sarcoma according to the U.S. Centers for Disease Control and Prevention Classification System for HIV-1 Infection within the past 12 months .
3. Any documented CD4+ T cell count < 200 cells/mm3 within the past 12 weeks .
4. Any exposure to a monoclonal antibody within the past 12 weeks.
5. Any significant diseases (other than HIV-1 infection) or clinically significant findings, that, in the Investigator's opinion, would preclude the subject from well participation or confound the assessment of study objectives.
6. Current receiving treatment regimen for Diabetes, hepatitis B, hepatitis C, or latent tuberculosis.
7. History of anaphylaxis to any monoclonal antibodies or HDAC inhibitor agents.
8. Received blood transfusion or hematopoietic growth factor treatment, any vaccine, or a compound with HDAC inhibitor activity (such as valproic acid) recently.
9. Use of immunomodulators, HIV vaccine, or systemic chemotherapy within 180 days prior to V1.
10. More than one change of ART regimen because of the inability to achieve or maintain suppression of viral replication to an HIV-1 RNA level < 200 copies/mL within the past 12 months
11. Receipt of any other investigational study agent(s) within 90 days.
12. Experienced urticaria in recent 6 months or ongoing or unresolved skin problems with rash-like symptoms .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
HIV-1 Total DNA levels | Post-treatment weeks up to 48 weeks
  The change in HIV-1 Total DNA from baseline after the study drug administration.

SECONDARY OUTCOMES:
HIV-1 Total DNA levels | Post-treatment weeks up to 48 weeks
  The changes in HIV-1 Total DNA levels during the study
Treatment related TEAE | through study completion, an average of 0.5 year
  The incidence of Grade 3 or higher grade drug-related treatment-emergent adverse events (TEAE)
Viral suppression | Post-treatment weeks up to 48 weeks
  Descriptive analysis of loss of viral suppression (HIV-1 VL> 50 copies/ml) during the study period.
The number of adverse subjects | Post-treatment weeks up to 48 weeks
  The number of adverse subjects leading to discontinuation of UB 421 or Chidamide.

CONTACTS AND LOCATIONS:
Overall Officials: undergoing undergoing, MD, Study Chair — undergoing